CLINICAL TRIAL: NCT01557270
Title: The Efficacy and Safety of Dexmedetomidine as an Additive to Ropivacaine for Interscalene Brachial Plexus Blocks for Shoulder Surgery
Brief Title: Efficacy and Safety Study of Dexmedetomidine as an Additive to Local Anesthetics in Shoulder Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Prof. Peter Gerner, M.D. (Other)
Responsible Party: Sponsor-Investigator, Prof. Peter Gerner, M.D., Professor, Paracelsus Medical University
Organization: Paracelsus Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GernerDex001
Record Dates: First submitted 2011-12-05; First posted 2012-03-19 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-12

CONDITIONS: Drug Safety; Self Efficacy
MeSH Terms: interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ropivacaine + dexmedetomidine (Experimental): This group represents the standard of care drug (ropivacaine) plus the new additive to be studied (dexmedetomidine)
  Interventions: Drug: dexmedetomidine
- ropivacaine + saline (Active Comparator): This group represents the current standard of care in peripheral nerve blockade
  Interventions: Drug: saline

INTERVENTIONS:
Drug: dexmedetomidine — ropivacaine 100 mg + 150 mcg dexmedetomidine, single shot perineural application
  Arms: ropivacaine + dexmedetomidine
Drug: saline — ropivacaine + saline placebo, single shot perineural application
  Arms: ropivacaine + saline

SUMMARY:
The purpose of this study is to test the efficacy and safety of dexmedetomidine added to ropivacaine in patients undergoing shoulder surgery.

DETAILED DESCRIPTION:
Peripheral nerve blocks are used throughout the world in lieu of general anesthesia and, more commonly, to provide analgesia and opioid sparing in the postoperative course. Long acting local anesthetics, such as ropivacaine, can provide analgesia for 11.5 ± 5 hours. This leads to many patients reporting their first pain in the evening and nighttime hours when access to healthcare providers and support is most limited. A number of additives to local anesthetics have been studied in humans with limited success. Recent work by a group in Michigan found a dose dependent increase in the duration of analgesia to a thermal stimulus when dexmedetomidine was added to ropivacaine for sciatic nerve blocks in rat.

The goal of the study is to investigate the safety and efficacy of dexmedetomidine added to ropivacaine for interscalene brachial plexus nerve block for shoulder surgery in humans. Provided the initial safety can be established, the trial will continue to evaluate secondary goals including the duration of analgesia, onset of sensory and motor blockade, and opioid-induced side effects. Tertiary outcomes will include subject satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III adult subjects
* Age 18-75
* Elective shoulder surgery
* Plan for interscalene brachial plexus block combined with general anesthesia
* Interscalene block
* Willingness to be contacted postoperatively for brief (5-10min) phone call questionnaires
* Written informed consent

Exclusion Criteria:

* Age < 18
* Age > 75
* Inability to understand protocol due to language barrier; difficulty with German language
* Chronic pain requiring daily opioids > 15 mg oral morphine equivalents (equals oral usage of > 10 mg oxycodone/daily; > 5 mg methadone/day; > 4 mg hydromorphone/day)
* Moderate (NRS pain score > 5) daily average pain
* Daily use of gabapentin, pregabalin, tricyclic antidepressant, serotonin- norepinephrine reuptake inhibitor, tramadol
* Hypersensitivity to amide local anesthetics
* History of hypersensitivity or allergic reaction to clonidine or dexmedetomidine
* Uncontrolled anxiety
* Schizophrenia or bipolar disorder
* Preexisting nerve damage (sensory or motor) in the extremity to be blocked
* Peripheral neuropathy
* Significant cardiovascular disease (second (Mobitz II type) or third degree heart block, congestive heart failure, chronic heart failure NYHA III-IV, symptomatic coronary artery disease CSS III-IV)
* BMI > 35
* Uncontrolled diabetes (blood sugar > 250 recorded in last 30 days or HbA1c > 7.5%)
* Chronic clonidine therapy (clonidine patch - Catapres or clonidine tablets)
* Hepatic Impairment (CHILD B or higher)
* Renal Impairment (creatinin > 2.0 mg/dl)
* Ongoing drug or alcohol abuse
* Pregnancy
* Prisoners

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2012-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Efficacy of dexmedetomidine in perineural application | 24 hrs
  The time until the patient describes the blockade as completely gone will be analysed and compared between the groups.
Safety of dexmedetomidine in perineural application | 30 days
  Any serious and/or unexpected adverse (AE) events will be assessed on an individual basis by the Principal Investigator and the DSMB. After the first twenty subjects (10 controls and 10 receiving study agent) have completed the study, the data will be reviewed. Provided the DSMB determines the initial safety is established, enrollment will proceed until a total of 62 subjects (31 subjects/group) have been accrued.

SECONDARY OUTCOMES:
Analgesia | first 24-48 hrs
  Analgesia will be assessed based on postoperative pain scores
Onset of sensory blockade | every 3 minutes for the first 21 minutes
  The subject's sensory function will be measured every 2 minutes for the first 20 minutes, until the loss of sensory function in the dermal distribution of the shoulder.
Duration of motor blockade | first 24-48 hrs
  The time to return of motor strength will be recorded in the subject's postoperative course.
Opioid-induced side effects | first 24-48 hrs
  Opioid-induced side effects will be recorded in the subject's postoperative course.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Gerner, MD, Principal Investigator — Paracelsus Medical University Salzburg, Department of Anesthesiology
Locations (1):
- Paracelsus Medical University, Department of Anesthesiology, Perioperative and Intensive Care Medicine, Salzburg, Austria

REFERENCES:
- [Background] Brummett CM, Amodeo FS, Janda AM, Padda AK, Lydic R. Perineural dexmedetomidine provides an increased duration of analgesia to a thermal stimulus when compared with a systemic control in a rat sciatic nerve block. Reg Anesth Pain Med. 2010 Sep-Oct;35(5):427-31. doi: 10.1097/AAP.0b013e3181ef4cf0. PMID 20814283
- [Background] Brummett CM, Hong EK, Janda AM, Amodeo FS, Lydic R. Perineural dexmedetomidine added to ropivacaine for sciatic nerve block in rats prolongs the duration of analgesia by blocking the hyperpolarization-activated cation current. Anesthesiology. 2011 Oct;115(4):836-43. doi: 10.1097/ALN.0b013e318221fcc9. PMID 21666435
- [Background] Brummett CM, Padda AK, Amodeo FS, Welch KB, Lydic R. Perineural dexmedetomidine added to ropivacaine causes a dose-dependent increase in the duration of thermal antinociception in sciatic nerve block in rat. Anesthesiology. 2009 Nov;111(5):1111-9. doi: 10.1097/ALN.0b013e3181bbcc26. PMID 19858875